CLINICAL TRIAL: NCT06260917
Title: The Effect of Urinating Through The Zipper or By Pulling Down The Trousers on Uroflowmetry Parameters in Patients With LUTS
Brief Title: The Effect of Urinating Through the Zipper or by Pulling Down the Trousers on Uroflowmetry Parameters in LUTS
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Turgay kacan, Principal investigator, Ankara City Hospital Bilkent
Other Study IDs: E2-23-4148
Record Dates: First submitted 2024-02-06; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Benign Prostatic Hyperplasia; Micturition Disorder; Urinary Obstruction; Urinary Tract Disease; Urologic Diseases
Keywords: benign prostatic obstruction; uroflowmetry; urodynamics
MeSH Terms: conditions — Prostatic Hyperplasia; Urination Disorders; Urologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- urination through zipper
  Interventions: Diagnostic Test: position of urination
- urinating by pulling down trousers
  Interventions: Diagnostic Test: position of urination

INTERVENTIONS:
Diagnostic Test: position of urination — effect of position on uroflowmetry parameters

SUMMARY:
There are many factors that affect uroflowmetry parameters. One of these is the urination position. Research has mostly focused on standing and sitting urination positions. However, those who prefer the standing position as a habit can urinate by opening the zipper or lowering the trousers. Although the effect of these two applications on uroflowmetry parameters in healthy men has been investigated in only one study, their effect on patients with lower urinary tract symptoms has not been examined.

ELIGIBILITY:
Inclusion Criteria:

* Having lower urinary tract symptoms due to BPO

Exclusion Criteria:

* Having a neurogenic bladder
* Previous prostate surgery
* Having urethral stricture
* Bladder neck stenosis
* Having a bladder stone or tumor
* Having a urinary system infection
* Finding a suspicious nodule in digital rectal examination

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on alpha blocker therapy with LUTS due to BPO
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Qmax | During the procedure
PVR | Immediately after procedure
Qave | During the procedure
Duration of voiding | During the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided